CLINICAL TRIAL: NCT04795336
Title: Melatonin Use After Primary Total Joint Arthroplasty: A Randomized, Double Blind Placebo-Controlled Trial
Brief Title: Melatonin Use After Primary Total Joint Arthroplasty
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-02030
Record Dates: First submitted 2021-03-05; First posted 2021-03-12 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Osteo Arthritis Knee
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Knee cohort (Active Comparator): In the cohort of patients undergoing primary elective knee arthroplasty, participants are recruited from those who are willing to consent and participate in the study, and will be randomly recruited into intervention group. Intervention group will receive a 5mg Melatonin prescription for 14 days
  Interventions: Drug: Melatonin 5 mg
- Knee cohort control (Placebo Comparator): In the cohort of patients undergoing primary elective knee arthroplasty, participants are recruited from those who are willing to consent and participate in the study, and will be randomly recruited into placebo group. Control group will receive a placebo pill for 14 days
  Interventions: Other: Placebo
- Hip cohort (Active Comparator): In the cohort of patients undergoing primary elective total hip, participants are recruited from those who are willing to consent and participate in the study, and will be randomly recruited into intervention group. Intervention group will receive a 5mg Melatonin prescription for 14 days
  Interventions: Drug: Melatonin 5 mg
- Hip cohort control (Placebo Comparator): In the cohort of patients undergoing primary elective total hip, participants are recruited from those who are willing to consent and participate in the study, and will be randomly recruited into placebo group. Control group will receive a placebo pill for 14 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Melatonin 5 mg — Melatonin is a widely sold synthetic molecule in various forms including tablets, gummies and liquid. In the present study, the tablet version of the medication will be used at a dose of 5mg
  Arms: Hip cohort; Knee cohort
Other: Placebo — The placebo ingredients are Microcrystalline Cellulose, Silica, Gelatin, Titanium Dioxide, Red #3, and Blue #1.
  Arms: Hip cohort control; Knee cohort control

SUMMARY:
The purpose of this study is to determine the effect of melatonin supplementation on patient sleep quality, length of stay, and opioid consumption following primary, unilateral, elective total hip or knee arthroplasty.

DETAILED DESCRIPTION:
This will be a single-center randomized double blind placebo control clinical trial. In the cohort of patients undergoing primary elective total hip and the cohort of patients undergoing primary elective knee arthroplasty, participants are recruited from those who are willing to consent and participate in the study, and will be randomly 1:1 divided into intervention group and placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Patient are current candidates for elective primary total hip and total knee arthroplasty.
* Patients ≥18 years of age but ≤ 95
* Patients have been medically cleared and scheduled for surgery

Exclusion Criteria:

* Non-elective conversion arthroplasty
* Bilateral total joint arthroplasty
* Contraindications to use of melatonin (diabetes, calcium channel blocker use, depression)
* Conditions and medications likely to confound results due to impact on subjective and/or objective sleep quality (insomnia, drug/alcohol abuse, and use of benzodiazepines, and prescription sleep aids)
* Conditions likely to impair capacity to adhere to protocol (mental impairment, psychiatric disorders other than anxiety/depression)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua C Rozell, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research. The investigator who proposed to use the data.
Access Criteria: Upon reasonable request. Requests should be directed to Daniel.waren@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Knee Cohort | Knee Cohort Control | Hip Cohort | Hip Cohort Control
Started | 69 | 69 | 78 | 78
Completed | 64 | 64 | 75 | 64
Not Completed | 5 | 5 | 3 | 14
Not completed — Withdrawal by Subject | 3 | 4 | 3 | 12
Not completed — Lost study logs | 0 | 1 | 0 | 2
Not completed — Did not take study medication | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Knee Cohort | Knee Cohort Control | Hip Cohort | Hip Cohort Control | Total
Number analyzed (Participants) | 64 | 64 | 75 | 64 | 267
Age, Continuous [Mean (Full Range); unit: years] | 64.1 [32 to 84] | 67.6 [41 to 83] | 62.7 [32 to 85] | 62.6 [24 to 83] | 63.9 [24 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 41 | 48 | 40 | 177
  Male | 16 | 23 | 27 | 24 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 3 | 5 | 8
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 64 | 64 | 72 | 59 | 259
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 1 | 5 | 3 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 14 | 13 | 10 | 6 | 43
  White | 43 | 38 | 54 | 46 | 181
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 12 | 6 | 9 | 30
Region of Enrollment [Number; unit: participants]
  United States | 64 | 64 | 75 | 64 | 267

OUTCOME MEASURES:

1. Primary Outcome: Change in Sleep Disturbance as Measured by Epworth Sleep Score (ESS)
Description: The primary objective is the Epworth Sleep Score used to evaluate the impact of melatonin use on the quality of sleep, including total hours of sleep and nighttime awakenings in patients undergoing elective primary total hip and knee arthroplasty. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.
Time Frame: Visit 1 (Screening Visit), Visit 2 (2 months post surgery)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Knee Cohort | Knee Cohort Control | Hip Cohort | Hip Cohort Control
Number analyzed (Participants) | 64 | 64 | 75 | 64
score on a scale | 7.2 (4.4) | 6.2 (4.1) | 6 (4) | 6.8 (4.5)

2. Secondary Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Score
Description: The PROMIS Sleep Disturbance questionnaire comprises 8 items assessing patients' sleep over the past 7 days. Each item is rated on a Likert scale from 1-5. The raw score is the sum of responses and is transformed to a normalized score from 0-100; higher scores indicate greater sleep disturbance.
Time Frame: Visit 1 (Screening Visit), 14 days after surgery visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Knee Cohort | Knee Cohort Control | Hip Cohort | Hip Cohort Control
Number analyzed (Participants) | 64 | 64 | 75 | 64
score on a scale | 4.6 (8.2) | 4 (8.4) | 0.3 (9.8) | 2.1 (9.8)

ADVERSE EVENTS:
Time Frame: 2 months
Description: Team monitored for adverse events at each study visit.
Arm/Group | Knee Cohort | Knee Cohort Control | Hip Cohort | Hip Cohort Control
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/64 | 0/75 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/64 | 0/75 | 0/64
Other Adverse Events (participants affected / at risk) | 0/64 | 0/64 | 0/75 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT04795336/Prot_SAP_000.pdf